CLINICAL TRIAL: NCT06378905
Title: Cukurova Score Validation Study in Prediction of Primary Cytoreduction in Advanced Ovarian Cancer
Brief Title: Cukurova Score Validation Study
Acronym: CUKUROVA
Status: Recruiting | Type: Observational
Sponsor: Cukurova University (Other)
Collaborators: Muğla Sıtkı Koçman University (Other); Sakarya University (Other); Gazi University (Other); Ankara Etlik City Hospital (Other Government); Kayseri City Hospital (Other Government); Mersin University (Other); Selcuk University (Other); Bezmialem Vakif University (Other); Uludag University (Other); Mersin City Hospital (Unknown); Marmara University (Other); Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other); Ankara University (Other); Ege University (Other); Hacettepe University (Other); Akdeniz University (Other); Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other); Mustafa Kemal University (Other); Trakya University (Other)
Responsible Party: Principal Investigator, Ghanim Khatib, Associate Professor, Cukurova University
Other Study IDs: 141/57
Record Dates: First submitted 2024-04-02; First posted 2024-04-23 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Epithelial Ovarian Cancer; Primary Cytoreduction
Keywords: Epithelial Ovarian Cancer; Cytoreduction
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite significant advancements in imaging technologies, surgical techniques, chemotherapeutic regimens, and treatment strategies in recent years, ovarian cancer continues to remain the most deadly gynecological malignancy. Approximately 90% of ovarian cancers originate from the coelomic epithelium or modified mesothelial cells and are classified as epithelial ovarian cancers. The majority of patients with epithelial ovarian cancer (70-80%) present in advanced stages. The primary treatment for advanced-stage (stage 3-4) disease consists of primary cytoreductive surgery followed by adjuvant chemotherapy. Cytoreductive surgery aims to remove all visible tumor implants regardless of the extent of the disease and achieve no visible residual tumor (complete cytoreduction, R0) at the end of the surgery. In cases where R0 cannot be achieved (due to poor general condition and/or extensive tumor that cannot be completely excised surgically), the option of neoadjuvant chemotherapy followed by interval cytoreductive surgery is considered. Primary cytoreductive surgery is still the preferred option and is considered a quality indicator for centers performing advanced-stage ovarian cancer surgeries. Despite advancements in surgery, the decision for interval surgery following primary surgery or neoadjuvant chemotherapy is often based on the surgeon's experience, imaging results, and clinic preferences. Various methods and scores have been published and applied to predict which patients are suitable for primary surgery.

The Cukurova score developed in our clinic conceptualizes prioritizing surgical procedures using radiological imaging and diagnostic exploratory laparoscopy to achieve complete cytoreduction in harmony with the patient's clinical and performance status, rather than focusing solely on tumor burden. The score showed high success rates for complete cytoreduction and also was useful in terms of predicting the morbidity and mortality. However, the Cukurova score study was conducted in single center. Validation of scores in centers with different capacities is expected to facilitate their widespread use and acceptance. Therefore, in this study, the investigators plan to conduct a validation study of the score in a total of 20 centers in Turkey, including our center. This study aims to evaluate the validity of the Cukurova score in predicting outcomes of primary cytoreduction in advanced ovarian cancer patients and thus determining the decision for primary cytoreductive surgery or neoadjuvant chemotherapy followed by interval cytoreductive surgery.

DETAILED DESCRIPTION:
Aim: The majority of patients with epithelial ovarian cancer (70-80%) present in advanced stages. The primary treatment for advanced-stage (stage 3-4) disease consists of primary cytoreductive surgery followed by adjuvant chemotherapy. Cytoreductive surgery aims to remove all visible tumor implants regardless of the extent of the disease and achieve no visible residual tumor (complete cytoreduction, R0) at the end of the surgery. In cases where R0 cannot be achieved (due to poor general condition and/or extensive tumor that cannot be completely excised surgically), the option of neoadjuvant chemotherapy followed by interval cytoreductive surgery is considered. Primary cytoreductive surgery is still the preferred option and is considered a quality indicator for centers performing advanced-stage ovarian cancer surgeries. Despite advancements in surgery, the decision for interval surgery following primary surgery or neoadjuvant chemotherapy is often based on the surgeon's experience, imaging results, and clinic preferences. Various methods and scores have been published and applied to predict which patients are suitable for primary surgery.

The Cukurova score developed in our clinic conceptualizes prioritizing surgical procedures using radiological imaging and diagnostic exploratory laparoscopy to achieve complete cytoreduction in harmony with the patient's clinical and performance status, rather than focusing solely on tumor burden. The score showed high success rates for complete cytoreduction and also was useful in terms of predicting the morbidity and mortality. However, the Cukurova score study was conducted in single center. Validation of scores in centers with different capacities is expected to facilitate their widespread use and acceptance. Therefore, in this study, the investigators plan to conduct a validation study of the score in a total of 20 centers in Turkey, including our center. This study aims to evaluate the validity of the Cukurova score in predicting outcomes of primary cytoreduction in advanced ovarian cancer patients and thus determining the decision for primary cytoreductive surgery or neoadjuvant chemotherapy followed by interval cytoreductive surgery.

Method: Informed consent forms will be obtained from all participants. Patients over the age of 18 suspected of having primary stage III-IV epithelial ovarian cancer will be included in this study. Cases with suspected peritoneal carcinomatosis findings on imaging studies or histologically confirmed at any time will be considered for the study. The followings are the exclusion criteria of the study; 1- refusing to participate in the study, 2- benign ovarian cases, 3- borderline ovarian tumors, 4- metastatic ovarian malignancies, 5- non-epithelial ovarian malignancies, 6- stage I-II epithelial ovarian cancers, and 7- being under 18 years old. Contrast-enhanced magnetic resonance imaging (MRI) will be preferred for abdominal imaging, and contrast-free computed tomography (CT) will be preferred for thoracic imaging. Imaging performed less than 3 weeks before surgery will be considered. Patients unable to undergo MRI will be evaluated with contrasted abdominopelvic CT scans. Imaging findings will be recorded, and necessary surgical procedures to achieve R0 will be discussed based on these findings, with a score assigned for each anticipated surgical procedure. These findings and anticipated surgical procedures are discussed through a multidiciplinary tumor board including at least two gynecological oncologists. Patients' age, body mass index, and performance scores will be recorded and scored, also. Scoring will be made according to the following parameters;

Each of 12 points:

* ECOG score ≥3
* ASA score ≥3
* Absolute stoma or blood transfusion refuse

Each of 2 points:

* Body mass index ≥40 or <18
* Age ≥75 years

Each of 12 points:

* Non-resectable extra-abdominal metastases
* Non-resectable multiple parenchymal liver metastases
* Non-resectable liver hilus involvement or non-repairable vessel-involved hepatoduodenal or celiac nodes
* Diffuse involvement of small bowel root represented in cocoon syndrome, non-movable or firmly retracted small bowel
* Confluent or extensive small bowel or meso involvement requiring resection which could lead to short bowel syndrome (<150cm)

Each of 6 points:

* Total gastrectomy
* Mesh necessitating diaphragmatic resection
* Ampullar region involvement requiring Whipple modifications
* Liver lobectomy
* Nephrectomy
* Total cystectomy
* Proctectomy

Each of 2 points:

* Liver segmentectomy (two points for each segment)
* Various surgical liver procedures (>2 procedures, covering >2 cm for each one, including metastasectomies, wedge resections, Glissonian excisions)
* Suprarenal lymphadenectomy(1)
* Splenectomy with or without distal pancreatectomy
* Bowel resections and anastomoses, 2 points for each anastomosis including small bowel anastomosis (eg, low anterior resection=2, total colectomy=2)
* Partial gastrectomy or full thickness gastric excisions
* Diaphragm stripping or primary sutured partial resections
* Ureteral anastomosis, 2 points for each one, including unilateral neocystostomy and significant partial cystectomy
* Video-assisted thoracic surgery (VATS)(2)

  1. Including direct suprarenal, hepatoduodenal, celiac, cardiophrenic, mediastinal, scalene, or cervical lymph nodes.
  2. Only in cases where surgical procedure is performed; diagnostic procedures with or without effusion drainage are not scored.

ASA, American Society of Anesthesiologists; ECOG, Eastern Cooperative Oncology Group.;

To calculate the clinic-Cukurova score; existing parameters' points are summed and multiplied by the ECOG score. In case of ECOG 0, only the summing process is done. Then diagnostic explorative laparoscopy ± VATS is performed and the required surgical procedures to achieve R0 are modified according to both radiological and laparoscopic evaluations. Again, the abovementioned parameters are scored and now the Cukurova score is calculated in similar manner (existing parameters' points are summed and multiplied by the ECOG score). Subsequently, in cases where the Cukurova score is equal or less than 12, primary debulking surgery will be performed. Neoadjuvant chemotherapy will be the choice in cases with Cukurova score more than 12. Laparoscopic evaluations will be approved by two gynecologic oncologists, and the decision regarding primary debulking surgery or neoadjuvant chemotherapy will be made with their agreement. If laparoscopic evaluation is inadequate due to extensive tumor adhesions and/or a large mass, Cukurova score will be calculated with a diagnostic explorative laparotomy. VATS will be performed in patients with pleural effusion and/or suspicious radiological findings in the thorax. Clinical, surgical, and postoperative follow-up information of the patients will be collected. Data collected from all centers will be statistically analyzed.

Sample size: According to the figures obtained from the Cukurova Score study, it has been observed that the R0 resection rate after primary debulking is 89%. Under the assumption that the AUC value for the Cukurova score in this group is 0.810, it has been calculated that at least 91 patients need to undergo primary debulking surgery with a 5% error rate and 90% power. Furthermore, considering that the percentage of patients undergoing primary debulking in this study is 70%, it has been planned to include at least 130 patients in total (including interval debulking patients).

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* Suspected advanced ovarian/fallopian tube/ primary peritoneal carcinomatosis on imaging
* Pathologically confirmed Stage III-IV epithelial ovarian cancer/fallopian tube/ primary peritoneal carcinomatosis
* Consent to participate in the study

Exclusion Criteria:

* Stage I-II epithelial ovarian/fallopian tube/peritoneal cancer
* Nonepithelial Ovarian Cancer
* Benign Ovarian tumors
* Borderline Ovarian Tumors
* Metastatic Ovarian Tumors
* Rejecting to Participate in the Study
* <18 years old

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women who have advanced epithelial ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Rate of complete cytoreduction | 1-3 years
  Complete cytoreduction (R0) is described as no visible residual tumor at the end of the surgery. The primary outcome of this study is to determine the rate of cases resulted with complete cytorection (R0).

SECONDARY OUTCOMES:
Rate of postoperative 90-days mortality | postoperative 90 days during the study period
  Rate of cases died during 90 days after surgery

OTHER OUTCOMES:
Rate of postoperative morbidity | postoperative 28 days during the study period
  Rate of grade 3 and more morbidity according to Dindo-Clavien classification.
  Grade-1:Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions.
  Grade-2:Requiring pharmacological treatment with drugs other than such allowed for Grade I complications. Blood transfusions and total parenteral nutrition (TPN) are also included.
  Grade-3:Requiring surgical, endoscopic or radiological intervention.
  Grade-4:Life-threatening complication (including those affecting the brain) requiring intensive care management.
  Grade-5:Death of a patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Khatib G, Seyfettinoglu S, Kose S, Kucukgoz Gulec U, Avci A, Guzel AB, Unal I, Paydas S, Vardar MA. The Cukurova score in the prediction of primary cytoreduction in ovarian cancer. Int J Gynecol Cancer. 2024 Jan 5;34(1):122-130. doi: 10.1136/ijgc-2023-004736. PMID 37945055
- [Background] Greimel E, Kristensen GB, van der Burg ME, Coronado P, Rustin G, del Rio AS, Reed NS, Nordal RR, Coens C, Vergote I; European Organization for Research and Treatment of Cancer - Gynaecological Cancer Group and NCIC Clinical Trials Group. Quality of life of advanced ovarian cancer patients in the randomized phase III study comparing primary debulking surgery versus neo-adjuvant chemotherapy. Gynecol Oncol. 2013 Nov;131(2):437-44. doi: 10.1016/j.ygyno.2013.08.014. Epub 2013 Aug 27. PMID 23994107
- [Background] Kehoe S, Hook J, Nankivell M, Jayson GC, Kitchener H, Lopes T, Luesley D, Perren T, Bannoo S, Mascarenhas M, Dobbs S, Essapen S, Twigg J, Herod J, McCluggage G, Parmar M, Swart AM. Primary chemotherapy versus primary surgery for newly diagnosed advanced ovarian cancer (CHORUS): an open-label, randomised, controlled, non-inferiority trial. Lancet. 2015 Jul 18;386(9990):249-57. doi: 10.1016/S0140-6736(14)62223-6. Epub 2015 May 19. PMID 26002111
- [Background] Fagotti A, Ferrandina G, Vizzielli G, Fanfani F, Gallotta V, Chiantera V, Costantini B, Margariti PA, Gueli Alletti S, Cosentino F, Tortorella L, Scambia G. Phase III randomised clinical trial comparing primary surgery versus neoadjuvant chemotherapy in advanced epithelial ovarian cancer with high tumour load (SCORPION trial): Final analysis of peri-operative outcome. Eur J Cancer. 2016 May;59:22-33. doi: 10.1016/j.ejca.2016.01.017. Epub 2016 Mar 19. PMID 26998845